CLINICAL TRIAL: NCT03616600
Title: The Safety and Effectiveness of Clinical Performance of Breath-O Correct Orthokeratology Lenses
Brief Title: The Safety and Effectiveness of Breath-O Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: SEED Co. Ltd. (Unknown)
Responsible Party: Principal Investigator, Henry HL Chan, PhD, Assocaite Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HongKongPU_Optometry2
Record Dates: First submitted 2018-03-15; First posted 2018-08-06 (Actual); Results first posted 2020-04-13 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-01

CONDITIONS: Myopia; Safety Issues
Keywords: Myopia; Orthokeratology
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Wearing the orthokeratology lenses for 3 months
  Interventions: Other: Breath-O-Correct Lens
- Control (No Intervention): Not wearing any contact lenses

INTERVENTIONS:
Other: Breath-O-Correct Lens — Breath-O correct lenses are new designed ready-made orthokeratology lenses which are made of new material with more elasticity as compared traditional lens material
  Arms: Treatment

SUMMARY:
In Hong Kong, approximately 80% of children are myopic by the end of childhood. There is intense interest currently in the potential role of peripheral defocus as a clinical treatment to slow myopia progression. One of the most successful treatments for myopia is orthokeratology. Currently, Breath-O correct lenses are new designed ready-made orthokeratology lenses. This study is to evaluate the safety of wearing this new orthokeratology lens and the effectiveness of clinical performance in young adult.

DETAILED DESCRIPTION:
Short-sightedness (myopia) is the most common refractive error in the world. In Hong Kong, approximately 80% of children are myopic by the end of childhood. Current treatment strategies to control (i.e. slow) myopia progression in children are primarily designed to harness the natural "emmetropization" process, in which visual feedback from retinal image clarity regulates the rate of eye growth. There is intense interest currently in the potential role of peripheral defocus as a clinical treatment to slow myopia progression, not least since this approach permits clear central vision. One of the most successful treatments for myopia is orthokeratology, which is a therapy of using custom-made rigid gas permeable contact lens. The special design of this contact lens can reshape the corneal profile to minimize the central refractive error while producing beneficial peripheral defocus. Currently, Breath-O correct lenses are new designed ready-made orthokeratology lenses which are made of new material with more elasticity as compared traditional lens material. This study is to evaluate the safety of wearing this new orthokeratology lens and the effectiveness of clinical performance in young adult.

ELIGIBILITY:
Inclusion Criteria:

1. Refractive error: Spherical: normally -1.00D to -4.00D (maximum up to -5.00D); Cylindrical: normally half of Sph (against-the-rule Astigmatism.: lower than -0.75D) (maximum up to -1.50D)
2. Best corrected Visual acuity: monocular ETDRS 0.0 or better
3. Ocular health: No ocular abnormality, no contra-indications for overnight orthokeratology lens wear, no refractive surgery
4. General health: No systemic diseases
5. Requirement: No history of orthokeratology lens wearing. Agree to participate in this study and willing to wear the orthokeratology lenses overnight in accordance with the instructions given and to come back for follow up within the study period

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-01-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 16 | 15
Completed | 15 | 15
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.8 (0.7) | 22.2 (2.4) | 21.1 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 4 | 6 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hong Kong | 15 | 15 | 30
Refractive errors [Mean (Standard Deviation); unit: Diopters] | -3.47 (1.01) | -3.71 (1.76) | -3.61 (1.40)

OUTCOME MEASURES:

1. Primary Outcome: Corneal Biomechanics in Terms of Corneal Hysteresis and Resistance Factor
Description: measured by ocular response analyser
Time Frame: Baseline, 1st Month, 3rd Month
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Treatment: Group randomly selected to wear the Breath-O Correct lenses
  Breath-O-Correct Lens: Breath-O correct lenses are new designed ready-made orthokeratology lenses which are made of new material with more elasticity as compared traditional lens material
- Control: Group randomly selected not to wear any contact lenses
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
mmHg
  Corneal Hysteresis_Baseline | 11.12 (1.12) | 11.10 (1.36)
  Corneal Hysteresis_1st Month | 10.37 (1.36) | 11.20 (1.89)
  Corneal Hysteresis_3rd Month | 10.14 (0.89) | 11.19 (1.66)
  Corneal Resistance Factor_Baseline | 11.07 (1.32) | 11.14 (2.23)
  Corneal Resistance Factor_1st Month | 9.87 (1.45) | 10.92 (2.45)
  Corneal Resistance Factor_3rd Month | 9.99 (1.37) | 10.79 (2.17)

2. Primary Outcome: Corneal Endothelial Health in Terms of Endothelial Cell Density
Description: measured by specular microscope
Time Frame: Baseline, 1st Month, 3rd Month
Measure: Mean (Standard Deviation); unit: cell/mm^2
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
cell/mm^2
  Corneal Endothelial Cell Density_Baseline | 2909 (145.1) | 2861 (181.05)
  Corneal Endothelial Cell Density_1st month | 2923 (123.01) | 2818 (182.65)
  Corneal Endothelial Cell Density_3rd month | 2917 (157.34) | 2825 (177.80)

3. Secondary Outcome: Best Corrected Visual Acuity in Terms of High and Low Contrast
Description: The best corrected visual acuity was measured in LogMAR (Snellen 20/20 vision = 0.00 in LogMAR ; each readable letter add -0.02 to the score, the smaller the number i.e. more negative, the better visual acuity)
Time Frame: Baseline, 1st Month and the 3rd Month
Population: It is a comparison of visual performance before-and-after treatment and therefore only the best corrected visual acuity in treatment group in different time points were compared.
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Treatment: Group randomly selected to wear the Breath-O Correct lenses
Arm/Group | Treatment
Number analyzed (Participants) | 15
LogMAR
  High contrast VA_Baseline | -0.10 (0.06)
  High contrast VA_1st Month | -0.07 (0.08)
  High contrast VA_3rd Month | -0.08 (0.08)
  Low contrast VA_Basline | 0.08 (0.08)
  Low contrast VA_1st Month | 0.22 (0.14)
  Low contrast VA_3rd Month | 0.17 (0.13)

4. Secondary Outcome: Reduction of the Refractive Power After Wearing the Breath-O-correct Lens
Description: Refractive errors were determined by subjective refraction for treatment group (Breath-O correct lens wearer), the outcome was represented as mean spherical equivalent refraction with unit in diopter (SER, = 1/2 Cylindrical power + spherical power)
Time Frame: Baseline, 1st Week, 1st Month, 3rd Month
Population: It is a comparison of refractive errors before-and-after treatment and therefore only the refractive errors in treatment group in different time points were compared.
Measure: Mean (Standard Deviation); unit: Diopter
Arm/Group | Treatment
Number analyzed (Participants) | 15
Diopter
  Refractive errors_Baseline | -3.52 (1.02)
  Refractive errors_1st Week | -0.17 (0.99)
  Refractive errors_1st Month | -0.11 (0.92)
  Refractive errors_3rd Month | -0.03 (0.82)

5. Primary Outcome: Corneal Endothelial Health in Terms of Percentage of Variation in Cell Size
Description: measured by specular microscope
Time Frame: Baseline, 1st Month, 3rd Month
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
percentage
  Corneal Endothelial Cell Variance_Baseline | 28.68 (3.78) | 29.35 (3.66)
  Corneal Endothelial Cell Variance_1st month | 28.47 (3.51) | 29.00 (3.58)
  Corneal Endothelial Cell Variance_3rd month | 29.00 (6.53) | 30.01 (3.32)

6. Primary Outcome: Anterior Ocular Health in Terms of Limbal and Bulbar Redness
Description: measured by OCULUS Keratograph® 5M and graded by JENVIS redness grading system It is a scale of 0 to 4, the higher the score, the more redness the ocular surface manifests
Time Frame: Baseline, 1st Month, 3rd Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
units on a scale
  Bulbar redness_Baseline | 0.57 (0.18) | 0.58 (0.28)
  Bulbar redness_1st Month | 0.47 (0.19) | 0.52 (0.21)
  Bulbar redness_3rd Month | 0.54 (0.31) | 0.61 (0.27)
  Limbal redness_Baseline | 0.26 (0.19) | 0.29 (0.26)
  Limbal redness_1st Month | 0.23 (0.15) | 0.31 (0.21)
  Limbal redness_3rd Month | 0.27 (0.21) | 0.38 (0.28)

7. Primary Outcome: Anterior Ocular Surface Evaluation in Terms of Non-invasive Keratography Break-up Time (NIKBUT)
Description: measured by OCULUS Keratograph® 5M
Time Frame: Baseline, 1st Month, 3rd Month
Measure: Mean (Standard Deviation); unit: Second
Arm/Group | Treatment | Control
Number analyzed (Participants) | 15 | 15
Second
  NIKBUT_1st break_Baseline | 6.72 (3.96) | 9.92 (6.76)
  NIKBUT_1st break_1st Month | 9.13 (5.45) | 9.17 (5.63)
  NIKBUT_1st break_3rd Month | 9.83 (6.37) | 7.64 (4.97)
  NIKBUT_average_Baseline | 10.94 (4.15) | 13.24 (6.56)
  NIKBUT_average_1st Month | 12.42 (5.73) | 11.86 (5.99)
  NIKBUT_average_3rd Month | 12.07 (6.76) | 9.57 (5.02)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 1/16 | 0/15
OTHER ADVERSE EVENTS (reported when occurring in more than 3.33% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=16) | Control (N=15)
poor visual quality (Eye disorders) | 1 | 0 — symptoms like glare and reduction in contrast from orthokeratology wearing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT03616600/Prot_SAP_000.pdf